CLINICAL TRIAL: NCT02600429
Title: Phase 3, Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of RGN-259 Ophthalmic Solution for the Treatment of Neurotrophic Keratopathy: SEER-1
Brief Title: Assessment of the Safety and Efficacy Study of RGN-259 Ophthalmic Solutions for Neurotrophic Keratopathy : SEER-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: ReGenTree, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-NK-301
Record Dates: First submitted 2015-10-26; First posted 2015-11-09 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Neurotrophic Keratopathy
Keywords: Neurotrophic Keratopathy; NK

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RGN-259 (Experimental): It is a preservative-free, sterile eye drop solution containing Tβ4
  Interventions: Drug: RGN-259
- Placebo (Placebo Comparator): It is composed of the same excipients as RGN-259 but does not contain Tβ4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGN-259 — A preservative-free, sterile eye drop solution containing Tβ4 for direct instillation into affected eye(s), five times a day for 4 weeks.
  Other Names: Tβ4
  Arms: RGN-259
Drug: Placebo — It is composed of the same excipients as RGN-259 but does not contain Tβ4
  Other Names: Vehicle Control
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety and efficacy of RGN-259 Ophthalmic Solution compared to placebo for the treatment of NK.

DETAILED DESCRIPTION:
Neurotrophic keratopathy (NK) is a degenerative corneal disease that occurs as a result of partial or total impairment of trigeminal innervation. The resulting loss of corneal sensitivity (anesthesia) leads to a reduction in lacrimation and a decline in status, metabolism, and mitosis of corneal epithelial cells. Previous studies (physician-sponsored studies) used to treat to nine patients with NK, six of whom had discrete geographic, non-healing lesions, and three of whom had punctate lesions and the study result reported.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female of any race, at least 18 years of age
* Have provided verbal and written informed consent.
* Be able and willing to follow instructions, including participation in all study assessments and visits;
* Have stage 2 or 3 neurotrophic keratopathy in at least one eye If a female of childbearing potential, have a negative urine pregnancy test at Visit 1 and agree to use an adequate method of birth control throughout the study period.

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that in the opinion of the investigator may interfere with the study parameters;
* Have significant blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergy that requires treatment
* Have a lid function abnormality (ex. Lagophthalmos) which, in the opinion of the investigator, is the primary cause of the persistent epithelial defect;
* Be diagnosed with ongoing ocular infection (bacterial, viral or fungal) or active inflammation (e.g. follicular conjunctivitis) not related to NK
* Anticipate the use of fluoroquinolone-containing antibiotic eye drops during the study;
* Have used contact lenses (excluding therapeutic contact lenses) within 14 days prior to Visit 1 or anticipates use of contact lenses during the study period;
* Have an uncontrolled systemic disease that in the opinion of the investigator may interfere with the study parameters;
* Anticipate a change in immunosuppressive therapy during the course of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Hull Eye Center, Lancaster, California
  - Vision Institute, Colorado Springs, Colorado
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Insight Vision Group, Parker, Colorado
  - Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - Midwest Cornea Associates, LLC, Indianapolis, Indiana
  - Koffler Vision Group, Lexington, Kentucky
  - Richard Eiferman, MD, PSC, Louisville, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Central Maine Eye Care, Lewiston, Maine
  - Black Hills Regional Eye Institute, Rapid City, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened prior to randomization. And after confirmation of inclusion and exclusion criteria, all eligible subjects were randomized in a 2:1 ratio to receive 0.1% RGN-259 or placebo ophthalmic solution bilaterally, five times per day for 28 days. The study comprised of 7 visits over the course of approximately 6 weeks.
Period: Overall Study
Arm/Group | RGN-259 | Placebo
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Total: Total of all reporting groups
Arm/Group | RGN-259 | Placebo | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 0 | 7
  >=65 years | 3 | 8 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (15.58) | 72.5 (7.87) | 67.6 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 6 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Complete Healing at Day 29.
Description: Percentage of subjects achieving complete healing of the persistent epithelial defect as determined by corneal fluorescein staining at day 29 after first dosing.
Time Frame: 29 days after first dosing
Measure: Count of Participants; unit: Participants
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
Participants | 6 | 1

2. Secondary Outcome: Percentage of Subjects Achieving Complete Healing at 8, 15, 22, 36, 43 Days
Description: Percentage of subjects achieving complete healing of the Persistent Epithelial Defect(PED) determined by corneal fluorescein staining at 8, 15, 22, 36, 43 days after first dosing.
Time Frame: 8, 15, 22, 36, 43 days after first dosing
Measure: Count of Participants; unit: Participants
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
Participants
  Percentage of subjects achieving complete healing of the PED at 8 days after first dosing. | 0 | 0
  Percentage of subjects achieving complete healing of the PED at 15 days | 3 | 1
  Percentage of subjects achieving complete healing of the PED at 22 days | 4 | 2
  Percentage of subjects achieving complete healing of the PED at 36 days | 4 | 1
  Percentage of subjects achieving complete healing of the PED at 43 days | 5 | 0

3. Secondary Outcome: Epithelial Defect Measurement and Classification as Stage 1, 2 or 3 Using Mackie Classification.
Description: Epithelial Defect Measurement and Classification as stage 1, 2 or 3 using Mackie Classification at 8, 15, 22, 29, 36, 43 days after first dosing
Time Frame: 8, 15, 22, 29, 36, 43 days after first dosing
Measure: Number; unit: participants
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
participants
  Epithelial Defect Measurement and Classification as stage 1 at 8 days after first dosing | 1 | 2
  Epithelial Defect Measurement and Classification as stage 2 at 8 days after first dosing | 8 | 6
  Epithelial Defect Measurement and Classification as stage 3 at 8 days after first dosing | 1 | 0
  Epithelial Defect Measurement and Classification as stage 1 at 15 days after first dosing | 4 | 3
  Epithelial Defect Measurement and Classification as stage 2 at 15 days after first dosing | 5 | 5
  Epithelial Defect Measurement and Classification as stage 3 at 15 days after first dosing | 0 | 0
  Epithelial Defect Measurement and Classification as stage 1 at 22 days after first dosing | 6 | 3
  Epithelial Defect Measurement and Classification as stage 2 at 22 days after first dosing | 3 | 5
  Epithelial Defect Measurement and Classification as stage 3 at 22 days after first dosing | 0 | 0
  Epithelial Defect Measurement and Classification as stage 1 at 29 days after first dosing | 6 | 2
  Epithelial Defect Measurement and Classification as stage 2 at 29 days after first dosing | 2 | 6
  Epithelial Defect Measurement and Classification as stage 3 at 29 days after first dosing | 0 | 0
  Epithelial Defect Measurement and Classification as stage 1 at 36 days after first dosing | 5 | 1
  Epithelial Defect Measurement and Classification as stage 2 at 36 days after first dosing | 3 | 6
  Epithelial Defect Measurement and Classification as stage 3 at 36 days after first dosing | 0 | 1
  Epithelial Defect Measurement and Classification as stage 1 at 43 days after first dosing | 4 | 1
  Epithelial Defect Measurement and Classification as stage 2 at 43 days after first dosing | 3 | 7
  Epithelial Defect Measurement and Classification as stage 3 at 43 days after first dosing | 0 | 0

4. Secondary Outcome: Tear Film Break-up Time at 29, 36, 43 Days
Description: Tear Film Break-up Time at 29, 36, 43 days after first dosing
Time Frame: 29, 36, 43 days after first dosing
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
Seconds
  Tear Film Break-up Time at 29 days after first dosing | 4.444 (3.3215) | 4.018 (2.8758)
  Tear Film Break-up Time at 36 days after first dosing | 4.131 (3.0701) | 3.658 (2.4115)
  Tear Film Break-up Time at 43 days after first dosing | 6.217 (6.7617) | 3.889 (2.1701)

5. Secondary Outcome: Ocular Discomfort by Questionnaire at 8, 15, 22, 29, 36, 43 Days After First Dosing
Description: Ocular Discomfort by Questionnaire at 8, 15, 22, 29, 36, 43 Days After First Dosing at Visits 2, 3, 4, 5, 6, and 7 (The scale used to determine the difference in Ocular Discomfort by questionnaire on each visit is from 0(None) to 5(Most). This outcome was calculated from two time points as the value at the later time point minus the value at the first dosing points and the lower value are considered to be a better outcome. and the all relevant time points used in the calculation in the Time Frame was 8, 15, 22, 29, 36, 43 days.)
Time Frame: 8, 15, 22, 29, 36, 43 days after first dosing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
score on a scale
  Ocular Discomfort by Questionnaire at 8 days after first dosing at Visits 2 | -1.5 (0.97) | -0.6 (1.19)
  Ocular Discomfort by Questionnaire at 15 days after first dosing at Visits 3 | -1.8 (0.79) | -0.3 (1.04)
  Ocular Discomfort by Questionnaire at 22 days after first dosing at Visits 4 | -1.7 (1.06) | -0.4 (0.92)
  Ocular Discomfort by Questionnaire at 29 days after first dosing at Visits 5 | -2.0 (1.05) | -0.3 (1.04)
  Ocular Discomfort by Questionnaire at36 days after first dosing at Visits 6 | -1.4 (1.43) | -0.1 (0.99)
  Ocular Discomfort by Questionnaire at 43 days after first dosing at Visits 7 | -1.4 (1.26) | -0.3 (1.28)

6. Secondary Outcome: Visual Acuity(logMAR) at 8, 15, 22, 29, 36, 43 Days
Description: Visual acuity(logMAR) at 8, 15, 22, 29, 36, 43 days
  (The Visual acuity was assessed by LogMAR calculation method. In the case of the LogMAR method, Each letter has a score value of 0.02 log units. Since there are 5 letters per line, the total score for a line on the LogMAR chart represents a change of 0.1 log units. and The lower value are considered to be a better outcome.)
  The formula used in calculating the score is:
  LogMAR VA = 0.1 + LogMAR value of the best line read - 0.02 X (number of optotypes read)
  used to determine the difference in Ocular Discomfort by questionnaire on each visit is the ORA scale: 0 None to 5: Most
  And as this outcome was calculated from two time points as the value at the later time point minus the value at the first dosing points, The lower value are considered to be a better outcome. and the all relevant time points used in the calculation in the Time Frame was 8, 15, 22, 29, 36, 43 days.)
Time Frame: 8, 15, 22, 29, 36, 43 days after first dosing
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
logMAR
  Visual acuity(logMAR) at 8 days | 1.451 (1.1873) | 1.090 (0.9697)
  Visual acuity(logMAR) at 15 days | 1.370 (1.3068) | 1.017 (1.0184)
  Visual acuity(logMAR) at 22 days | 1.287 (1.3616) | 1.020 (1.0097)
  Visual acuity(logMAR) at 29 days | 1.323 (1.3283) | 1.003 (1.0315)
  Visual acuity(logMAR) at 36 days | 1.280 (1.3542) | 0.990 (1.0315)
  Visual acuity(logMAR) at 43 days | 1.424 (1.4556) | 0.997 (1.0292)

7. Other Pre Specified Outcome: The Number of Participants With an Abnormal Findings by Slit-lamp Biomicroscopy at 8, 15, 22, 29, 36, 43 Days
Description: The number of participants with a abnormal findings by Slit-lamp biomicroscopy at 8, 15, 22, 29, 36, 43 days
  This outcome was assessed by the number of participants with an abnormal findings which are clinically significant using slit-lamp biomicroscopy which provides a magnified view of intraocular structures in the Cornea, Conjunctiva, Anterior Chamber, Iris, Lens, Eyelid.
Time Frame: 8, 15, 22, 29, 36, 43 days after first dosing
Measure: Number; unit: participants
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
participants
  Abnormal findings at 8 days | 6 | 5
  Abnormal findings at 15 days | 6 | 5
  Abnormal findings at 22 days | 6 | 5
  Abnormal findings at 29 days | 6 | 5
  Abnormal findings at 36 days | 7 | 5
  Abnormal findings at 43 days | 6 | 5

8. Other Pre Specified Outcome: Corneal Sensitivity Using the Aesthesiometer (Cochet-Bonnet)
Description: Corneal Sensitivity using the aesthesiometer (Cochet-Bonnet) at 29, 43 days after first dosing
Time Frame: 29, 43 days after first dosing
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
mm
  Corneal Sensitivity in Study Eye at 29 days | 11.77 (17.708) | 14.38 (17.336)
  Corneal Sensitivity in Study Eye at 43 days | 12.87 (16.648) | 18.33 (25.136)

9. Other Pre Specified Outcome: The Number of Participants With an Abnormal Findings by Dilated Fundoscopy at 29, 43 Days
Description: The number of participants with an abnormal findings by Dilated Fundoscopy at 29, 43 days
  This outcome was assessed by the number of participants with an abnormal findings which are clinically significant using Dilated Fundoscopy which is a diagnostic procedure to view the eye's interior, allowing assessment of the Vitreous, Retina, Macula, Choroid, and Optic Nerve.
Time Frame: 29, 43 days after first dosing
Measure: Number; unit: participants
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
participants
  Biomicroscopy in study eye at 29 days | 1 | 0
  Biomicroscopy in study eye at 43 days | 1 | 0

10. Other Pre Specified Outcome: Intraocular Pressure
Description: Intraocular Pressure at 29, 43 days after first dosing
Time Frame: 29, 43 days after first dosing
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RGN-259 | Placebo
Number analyzed (Participants) | 10 | 8
mmHg
  Intraocular Pressure in study eye at 29 days | 18.0 (6.60) | 14.5 (4.41)
  Intraocular Pressure in study eye at 43 days | 16.8 (6.23) | 12.5 (2.73)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at every visit through study completion, approximately 6 weeks.
Description: There was no anticipated/unanticipated deaths due to any cause in this study.
Arm/Group | RGN-259 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 4/10 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGN-259 (N=10) | Placebo (N=8)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGN-259 (N=10) | Placebo (N=8)
Corneal epithelium defect (Eye disorders) | 2 (2) | 0 (0)
Corneal opacity (Eye disorders) | 1 (2) | 0 (0)
Keratic precipitates (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (3)
Inflammation (General disorders) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Upper repiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT02600429/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT02600429/SAP_001.pdf